CLINICAL TRIAL: NCT06330038
Title: Recurrence Free Survival After Curative Resection of Non-small Cell Lung Cancer Between Inhalational Gas Anesthesia and Propofol-based Total IntraVenous Anesthesia: a Multicenter, Randomized, Clinical Trial
Brief Title: Anesthesia and Non-small Cell Lung Cancer Recurrence
Acronym: GASTIVA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Asan Medical Center (Other); Severance Hospital (Other); Seoul St. Mary's Hospital (Other); Korea University Guro Hospital (Other); DongGuk University (Other); Inha University Hospital (Other); Konkuk University Medical Center (Other); Ewha Womans University (Other); Chungnam National University Hospital (Other); University of Virginia (Other); Memorial Sloan Kettering Cancer Center (Other); Yale University (Other); Mayo Clinic (Other); University of Texas Southwestern Medical Center (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Khon Kaen University (Other); King Chulalongkorn Memorial Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Beijing Hospital (Other Government); All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SMC 2024-01-065
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer; Surgery; Anesthesia
Keywords: Anesthesia; Desflurane; Inhalational anesthesia; Isoflurane; Lung neoplasm; Metastasis; Propofol; Recurrence; Sevoflurane; Surgery; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Propofol; Sevoflurane; Desflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA group (Experimental): The TIVA group will receive propofol for both induction and maintenance of general anesthesia.
  Interventions: Drug: Propofol
- GAS group (Active Comparator): The GAS group will receive one or more volatile anesthetics (sevoflurane, desflurane, or isoflurane) for induction and maintenance of anesthesia during the surgery. For GAS group, propofol, midazolam, remimazolam, etomidate, or ketamine can be used with inhalation agents as co-induction agents under the discretion of the attending anesthesiologist.
  Interventions: Drug: Inhaled anesthetics

INTERVENTIONS:
Drug: Propofol — Propofol will be used for the induction and maintenance of general anesthesia.
  Other Names: Propofol 1% or 2% inj.
  Arms: TIVA group
Drug: Inhaled anesthetics — Inhaled anesthetics will be used for the maintenance of general anesthesia.
  Other Names: Sevoflurane, Desflurane, Isoflurane
  Arms: GAS group

SUMMARY:
There has been ongoing debate about the relationship between cancer recurrence and anesthetic management. Therefore, the investigators will test the hypothesis that the recurrence free survival (RFS) after curative resection of NSCLC is higher in patient who received total intravenous anesthesia (TIVA) than volatile anesthetics in this multi-center randomized trials.

DETAILED DESCRIPTION:
Surgery is the primary treatment for non-small cell lung cancer (NSCLC), but microscopic residual disease may be unavoidable. Preclinical studies have shown that volatile anesthetics might suppress host immunity and promote a pro-malignant environment which supports cancer cell proliferation, migration, and angiogenesis, whereas propofol may preserve cell-mediated immunity and inhibits tumor angiogenesis. However, clinical evidence that propofol-based total intravenous anesthesia (TIVA) can reduce tumor recurrence after curative resection remains inconsistent due to retrospective observational nature of previous studies. Therefore, the investigators will test the hypothesis that the recurrence free survival (RFS) after curative resection of NSCLC is higher in patient who received TIVA than volatile anesthetics in this multi-center randomized trials.

This double-blind, randomized trial will enroll patients at 22 international sites, subject to study registration, institutional review board approval, and patient written informed consent. Eligible patients are adult patients undergoing lung resection surgery with curative intent for NSCLC. At each study site, enrolled subjects will be randomly allocated into the TIVA and GAS group with a 1:1 ratio. A centralized, password-protected, and encrypted web-based electronic case report form will be used for randomization and data upload. This pragmatic trial does not standardize any aspect of patient care. However, potential confounders will be balanced between the study arms.

The primary outcome will be recurrence free survival (RFS). Secondary outcomes will be overall survival and complications within postoperative 7 days. Enrollment of 5384 patients will provide 80% power to detect a 3% treatment effect (hazard ratio of 0.83) at alpha 0.05 for RFS at 3 years.

Confirmation of the study hypothesis would demonstrate that a relatively minor and low cost alteration in anesthetic management has the potential to reduce cancer recurrence risk in NSCLC, an ultimately fatal complication. Rejection of the hypothesis would end the ongoing debate about the relationship between cancer recurrence and anesthetic management.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA) Ⅰ-Ⅲ
* The Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Lung resection surgery (segmentectomy, lobectomy, bilobectomy, pneumonectomy; video-assisted, robot-assisted, or open) with curative intent for NSCLC (clinical Tumor, Node, Metastasis (TNM) stage Ⅰ- ⅢA).

Exclusion Criteria:

* Distant metastasis or malignant tumor in other organs that according to the attending surgeon is not in long-term remission
* Severe neurologic conditions
* Severe hepatic disease (Child-Pugh classification C)
* Renal failure requiring renal replacement therapy
* History of anesthesia and/or surgery within 1 yr
* Previous surgery due to lung cancer (except diagnostic biopsies)
* Contraindications to any study medication (history of allergy, hypersensitivity reaction, or any other contraindication)
* Planned joint extrapulmonary procedure
* Surgery under cardiopulmonary bypass or extracorporeal membrane oxygenation
* Postoperative sedation
* Pregnancy, or lactation
* Patient refusal.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5384 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | Within 3 year after curative resection for NSCLC
  Time from surgery to the earliest date of local recurrence/metastasis or death from any cause, whichever comes first

SECONDARY OUTCOMES:
Overall survival | Within 3 year after curative resection for NSCLC
  Time from index surgery to death due to any causes
Postoperative complications | within 7 days post-surgery or at discharge if earlier
  Rate of complications which will be assessed with Clavien-Dindo classification and postoperative complications defined by the Society of Thoracic Surgeons (STS) general thoracic surgery databases

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, Principal Investigator — Department of Anesthesiology and Pain Medicine, Samsung Medical Center

IPD SHARING:
Plan to Share IPD: Yes
Data sharing including the full protocol, individual participant and other relevant study data will be considered upon reasonable request. Only with the permission of the Data Review Board of Samsung Medical Center, the anonymized data will be available from the principal investigator (HJA).
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: within 3 years after publication
Access Criteria: Data sharing including the full protocol, individual participant and other relevant study data will be considered upon reasonable request. Only with the permission of the Data Review Board of Samsung Medical Center, the anonymized data will be available from the principal investigator (HJA).

REFERENCES:
- [Derived] Kim J, Yoon S, Song IK, Lee K, Hwang W, Kim H, Lee DK, Lim HK, Kim SH, Lee JW, Hong B, Blank RS, Pedoto A, Popescu W, Theresa G, Martin AK, Patteril M, Pathanasethpong A, Thongsuk Y, Pisitpitayasaree T, Huang A, Yu H, Kapoor PM, Kim K, Chi SA, Ahn HJ. Recurrence-free survival after curative resection of non-small cell lung cancer between inhalational gas anesthesia and propofol-based total intravenous anesthesia: a multicenter, randomized, clinical trial (GAS TIVA trial): protocol description. Perioper Med (Lond). 2024 Jul 23;13(1):79. doi: 10.1186/s13741-024-00436-1. PMID 39039548